CLINICAL TRIAL: NCT05440188
Title: Identification of the Reduction of Exacerbations Resulting in Hospital Admission in COPD Patients After the Use of the Breath Detect Telemedicine Platform.
Brief Title: Study to Identify the Reduction of Exacerbations Resulting in Hospital Admission in Patients With COPD.
Acronym: BDS
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Principal Investigator, Universidad Autonoma de Madrid
Other Study IDs: Breath Detect Study
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: COPD Exacerbation
Keywords: telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD: Patients over 65 years old diagnosed with COPD in GOLD II state or higher who uses Breath Detect Platform for monitoring their respiratory health status.
  Interventions: Diagnostic Test: Breath Detect Platform

INTERVENTIONS:
Diagnostic Test: Breath Detect Platform — Use of the Breath Detect platform for respiratory health monitoring.

SUMMARY:
identification of the reduction of exacerbations resulting in hospital admission in COPD patients after the use of the Breath Detect telemedicine platform.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosed in GOLD II state or higher

Exclusion Criteria:

* Can´t read and talk in spanish

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients from Primary Health Care, Elderly care homes, and HULP
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Number of hospital admissions due to exacerbations | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CS Entrevías, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided